CLINICAL TRIAL: NCT04456543
Title: Comparison and Clinical Utility of the Portable Pressure Measuring Device for Garment Pressure Measurement on Hypertrophic Scar by Burn Injury During Compression Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HangangSHH-11
Record Dates: First submitted 2020-06-08; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Burns; Hypertrophic Scar
Keywords: burns; compression therapy; skin characteristics; hypertrophic scar; pressure sensor
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: patients with partial-/full-thickness burns, which spontaneously healed or required skin grafting, from the Department of Rehabilitation Medicine at the Hangang Sacred Heart Hospital of Korea
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are randomly devided into two groups. Outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure monitoring group (Experimental): In the pressure monitoring group, garment pressures were monitored using the portable pressure measuring device and the compression garment was adjusted so that the pressure was maintained at the therapeutic range of 15 - 25 mmHg for 2 months. Subjects were instructed to wear the garment 23 hours per day, removing them only for bathing.
  Interventions: Procedure: pressure monitoring
- conventional treatment group (Active Comparator): In the conventional treatment group, non-surgical standard treatment of burn scars except for pressure monitoring was performed in the same manner. Subjects were instructed to wear the garment 23 hours per day, removing them only for bathing.
  Interventions: Procedure: pressure monitoring

INTERVENTIONS:
Procedure: pressure monitoring — garment pressures were monitored using the portable pressure measuring device and the compression garment was adjusted so that the pressure was maintained at the therapeutic range of 15 - 25 mmHg.

SUMMARY:
The investigators developed a portable pressure measuring device using silicon piezoresistive pressure sensors. As PicoPress® is the most accurate (i.e., lowest variation and error) manometric sensor for pressure measurement, the investigators used it to compare and examine the accuracy of the proposed device regarding in vitro pressure measurements. The purpose of this study was to determine the effectiveness of pressure garment therapy using proposed device with objective data obtained with a randomized within wound comparison. Pressure measurements were acquired through a readout circuit consisting of an analog-to-digital converter, a microprocessor, and a Bluetooth transmission module for wireless data transmission to an external device. The mean pressure values measured by the sensors were compared to those obtained from PicoPress®. This was a double-blinded, randomized, controlled trial of patients with hypertrophic scars. In the pressure monitoring group, garment pressures were monitored using the portable pressure measuring device, and the compression garment was adjusted so that the pressure was maintained at the therapeutic range of 15 - 25 mmHg. In the control group, non-surgical standard treatment of burn scars except for pressure monitoring was performed in the same manner.

DETAILED DESCRIPTION:
The investigators developed a portable pressure measuring device using silicon piezoresistive pressure sensors. As PicoPress® is the most accurate (i.e., lowest variation and error) manometric sensor for pressure measurement, the investigators used it to compare and examine the accuracy of the proposed device regarding in vitro pressure measurements. The purpose of this study was to determine the effectiveness of pressure garment therapy using proposed device with objective data obtained with a randomized within wound comparison. Pressure measurements were acquired through a readout circuit consisting of an analog-to-digital converter, a microprocessor, and a Bluetooth transmission module for wireless data transmission to an external device. The mean pressure values measured by the sensors were compared to those obtained from PicoPress®. This was a double-blinded, randomized, controlled trial of patients with hypertrophic scars. In the pressure monitoring group, garment pressures were monitored using the portable pressure measuring device, and the compression garment was adjusted so that the pressure was maintained at the therapeutic range of 15 - 25 mmHg. In the control group, non-surgical standard treatment of burn scars except for pressure monitoring was performed in the same manner. To evaluate the effect of a pressure monitoring device, the investigators compared the skin test results (thickness, melanin, erythema, TEWL, and skin elasticity levels) between the two groups, from baseline measures immediately before the treatment and measures immediately after 2 months. The participants were made comfortable and acclimatized to room conditions. Room temperature was maintained at 20-25'C and relative humidity at 40-50 %. In the supine position, skin properties were measured. The thickness was measured with a ultrasonic wave equipment (128 BW1 Medison, Korea). Mexameter® (MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure melanin levels and the severity of erythema. The higher values indicating a darker and redder skin. Transepidermal water loss (TEWL) was measured with a Tewameter® (Courage-Khazaka Electronic GmbH, Germany), which is used for evaluating water evaporation. Elasticity was measured using Cutometer SEM 580® (Courage-Khazaka Electronic GmbH, Cologne, Germany), which applies negative pressure (450 mbar) on the skin. The numeric values (mm) of the skin's distortion is presented as the elasticity. Two seconds of negative pressure of 450 mbar is followed by 2 s of recess, and this consists of a complete cycle. Three measurement cycles were conducted, and the average values were obtained. The parameters consist of the following biomechanical skin properties: distenstibility, elasticity, and viscoelasticity. Distensibility means the length of total displacement from initial postion at maximum negative pressure. Gross elasticity means the ability of the skin to return to its initial position following displacement. Biologic elasticity means the ratio of immediate retraction to total displacement. Viscoelasticity means the ratio of delayed distension of immediate distension. Outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention. Possible complications (pain, ecchymosis, pain, skin abrasion, and swelling) were observed.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* partial-/full-thickness burns
* fully epithelialization after spontaneously healed or required skin grafting

Exclusion Criteria:

* open wounds
* infection on the burn scars
* those taking steroids for the scars
* condition affecting wound healing (e.g., diabetes)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline scar thickness at 8 weeks | 8 weeks (before intervention and 8 weeks after intervention)
  hypertrophic scar thickness. The thicker the measurement thickness, the larger the number.

SECONDARY OUTCOMES:
Change from baseline scar pigmentation at 8 weeks | 8 weeks (before intervention and 8 weeks after intervention)
  measurement of melanin level. The higher values indicating a darker
Change from baseline scar erythema at 8 weeks | 8 weeks (before intervention and 8 weeks after intervention)
  The higher values indicating a redder skin.
Change from baseline skin dryness at 8 weeks | 8 weeks (before intervention and 8 weeks after intervention)
  measurement of transepidermal water loss. The higher the measurement, the dryer the skin.
Change from baseline skin elasticity at 8 weeks | 8 weeks (before intervention and 8 weeks after intervention)
  Biologic elasticity means the ratio of immediate retraction to total displacement using suction. The higher the measurement, the more elasticity

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeongdeungpo-Ku, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harries CA, Pegg SP. Measuring pressure under burns pressure garments using the Oxford Pressure Monitor. Burns. 1989 Jun;15(3):187-9. doi: 10.1016/0305-4179(89)90180-0. PMID 2757769
- [Background] Li-Tsang CW, Zheng YP, Lau JC. A randomized clinical trial to study the effect of silicone gel dressing and pressure therapy on posttraumatic hypertrophic scars. J Burn Care Res. 2010 May-Jun;31(3):448-57. doi: 10.1097/BCR.0b013e3181db52a7. PMID 20375696
- [Background] Macintyre L, Baird M. Pressure garments for use in the treatment of hypertrophic scars--a review of the problems associated with their use. Burns. 2006 Feb;32(1):10-5. doi: 10.1016/j.burns.2004.06.018. PMID 16413399